CLINICAL TRIAL: NCT04454697
Title: Geweberetraktoren für Die Strahlentherapie Von Kopf-Hals-Tumoren - Prospektive Randomisierte Phase-II-Studie
Brief Title: Tissue Retractors for Radiation Therapy of Head and Neck Tumors
Acronym: GUARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUARD
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventiongroup: Personalized GWR Controlgroupt: standardized radiation protection tooth splints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patient receive personalized 3D-printed GWR
  Interventions: Device: tissue retractors
- Control (Active Comparator): Patient receive standardized radiation protection tooth splints
  Interventions: Device: tissue retractors

INTERVENTIONS:
Device: tissue retractors — Patients receive a tissue retractor to spare healthy tissue during the course of radiation

SUMMARY:
The rate of therapy-associated side effects during and after radiotherapy of head and neck tumors is essential. The most effective approach to reducing acute toxicity is to cut out healthy tissue from the radiation field. The distance between the tumor and normal tissue can be individually increased using personalized, 3D printer-based tissue retractors (GWR). Even the smallest geometric changes lead to a significant dose reduction in normal tissue and significant advantages for the patient.

The current randomized phase II study evaluates the use of GWR with regard to acute toxicity. In addition, quality of life, long-term toxicity as well as local control and overall survival 12 months after radiotherapy are evaluated.

DETAILED DESCRIPTION:
The most effective approach to reducing acute toxicity after radiotherapy is to cut out healthy tissue from the radiation field. GWR can increase the distance between the tumor and normal tissue. Even the smallest geometric changes lead to a significant dose reduction in normal tissue and significant advantages for the patient. Adequate immobilization also reduces unwanted movements, especially of the tongue.

The GWR are manufactured as combinable modules according to the "modular principle". This improves reproducibility and flexibility and reduces development and manufacturing costs. The study is being conducted as a monocentric, prospective, randomized phase II study. A total of 34 patients who meet the inclusion criteria are examined for acute toxicity after radiotherapy of a malignant head and neck tumor. The primary goal of the study is to reduce acute toxicity through individual immobilization of the jaw and tongue. Secondary study goals are the evaluation of quality of life and long-term toxicity as well as local control and overall survival twelve months after radiotherapy. In both groups, radiation therapy is carried out in accordance with guidelines using image-guided radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a malignant head and neck tumor
* Clinical target volume of radiotherapy may include portions of at least one region: oral cavity; Upper jaw; Lower jaw; Oropharynx; Hypopharynx; large salivary glands
* Indication for radiotherapy alone (postoperative or definitive)
* Age ≥ 18 years
* Karnofsky performance score ≥ 60
* Completed wound healing after tumor resection
* The patient's consent and written consent
* Ability of the patient to assess the nature and scope as well as possible consequences of the clinical study
* Adequate contraception in women of childbearing potential and in men

Exclusion Criteria:

* Pre-radiation in the head and neck area
* Multifocal, diffuse growing tumors
* Inadequate regression of toxicities from previous therapies
* Jaw clamp (cutting edge distance ≤ 2 cm)
* Simultaneous systemic tumor therapy during radiation (especially chemotherapy and immunotherapy)
* Indications that the participant is unlikely to adhere to the study protocol (e.g. lack of compliance)
* Missing written declaration of consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Toxcicity | immediately after completin of Radiotherapy
  Number of grade III toxcicity events

SECONDARY OUTCOMES:
Assesment of Quality of life: questionnaire | up to 12 month after completion of radiotherapy
  Changes of Parameters on the Core Quality of Life Questionnaire C30, scores 1 to 6 (best)
Assesment of Quality of life: questionnaire | up to 12 month after completion of radiotherapy
  Changes of Parameters on the Core Quality of Life Questionnaire H&N35, scores 1 to 6 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Adeberg, PD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hopsital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroter P, Christ LV, Dvornikovich K, Stritzke F, Franke H, Weusthof K, Bauer L, Regnery S, Deng M, Behnisch R, Kolz TT, Herpel C, Tholken R, Schuler P, Moratin J, Ristow O, Rammelsberg P, Hoffmann J, Schwindling FS, Uzun-Lang K, Herfarth K, Adeberg S, Debus J, Held T. Randomized controlled trial of semi-individualized 3D-printed tissue retraction devices vs. standard shielding splints in head and neck cancer treated with intensity-modulated and particle radiotherapy (GUARD). Oral Oncol. 2025 Oct;169:107604. doi: 10.1016/j.oraloncology.2025.107604. Epub 2025 Aug 20. PMID 40840174
- [Derived] Held T, Herpel C, Schwindling FS, Christ L, Lang K, Regnery S, Eichkorn T, Hommertgen A, Jaekel C, Krisam J, Moratin J, Mrosek J, Metzger K, Zaoui K, Moutsis T, Harrabi S, Herfarth K, Freudlsperger C, Rammelsberg P, Debus J, Adeberg S. 3D-printed individualized tooth-borne tissue retraction devices compared to conventional dental splints for head and neck cancer radiotherapy: a randomized controlled trial. Radiat Oncol. 2021 Apr 17;16(1):75. doi: 10.1186/s13014-021-01803-8. PMID 33865401